CLINICAL TRIAL: NCT00638638
Title: Myocardial Infarction With ST-elevation Treated by Primary Percutaneous Intervention Facilitated by Early Reopro Administration in Alsace.
Brief Title: Myocardial Infarction With ST-Elevation
Acronym: MISTRAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Christine GEILLER, directeur Adjoint, University Hospital, Strasbourg, France
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3233
Record Dates: First submitted 2008-02-28; First posted 2008-03-19 (Estimated); Last update posted 2009-09-17 (Estimated); Status verified 2009-09

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Angioplasty; Coronary stenting; Abciximab; Myocardial reperfusion; Microcirculation; EKG; ST elevation myocardial infarction within 6 h of symptom onset
MeSH Terms: conditions — Myocardial Infarction | interventions — Abciximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): * Early Abciximab bolus during prehospital transportation in ambulance 0.25 mg/Kg iv with Heparin 40 UI/kg bolus.
  * Abciximab placebo bolus and Abciximab infusion 10 µg/Kg/min after coronary angiography and before angioplasty.
  Interventions: Drug: Abciximab; Drug: Abciximab placebo
- 2 (Experimental): * Abciximab placebo bolus during prehospital transportation in ambulance with Heparin 40 UI/kg bolus.
  * Abciximab 0.25 mg/Kg bolus after coronary angiography and before angioplasty followed by Abciximab infusion 10 µg/Kg/min.
  Interventions: Drug: Abciximab; Drug: Abciximab placebo

INTERVENTIONS:
Drug: Abciximab — * Abciximab: 0.25 mg/Kg bolus
  * Abciximab placebo bolus
  * Abciximab infusion 10 µg/Kg/min
  Other Names: 1: Experimental; 2: Experimental
Drug: Abciximab placebo — * Abciximab placebo Bolus
  * Abciximab: 0.25 mg/Kg bolus
  * Abciximab infusion 10 µg/Kg/min
  Other Names: 1: Experimental; 2: Experimental

SUMMARY:
Mechanical recanalization of the culprit artery in acute myocardial infarction using stents provides in 2003, TIMI 3 flow restoration in more than 90% of patients. However, the prognosis of this condition remains poor, to a large degree because of microcirculatory dysfunction that is observed, in near than 20 to 40 % of patients, during or following primary percutaneous intervention. The lack of ST-segment elevation resolution after angioplasty with stenting is a marker of microcirculatory dysfunction and is associated with a poor prognosis. Routine administration with primary stenting of the platelet glycoprotein IIb/IIIa inhibitor Abciximab in acute myocardial infarction is still a matter of debate with conflicting results emerging from two major clinical studies ADMIRAL and CADILLAC. However, evidences are in favour of a benefit of this treatment especially when administrated early (in a pre-hospital manner) before percutaneous coronary intervention.Our primary purpose is to investigate the benefit of an early (i.e. pre-hospital) vs. a conventional (i.e. per-angiography) administration of Abciximab on ST-segment elevation regression at one hour after primary percutaneous angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age eligible for randomization in the MICU
* Infarct within 6 hours from symptoms onset
* Continuous typical chest pain symptoms symptoms for more than 20 min. and-ST segment elevation of more than 2 mm in more than two leads (peripheral or precordial)
* Signed informed consent form

Exclusion Criteria:

* Ventricular conduction anomalies masking signs of ischemia (left or right bundle branch block without evidence of additional elevation), electrical left ventricular hypertrophy
* Known hypersensitivity to Abciximab or to any component of the product or to murine monoclonal antibodies.- Hemorrhagic diathesis, internal hemorrhage
* Hemorrhagic stroke within 2 years
* Ischemic stroke within the last 3 months- Intra-cranial neoplasm, intracranial malformation or arteria
* venous aneurysm
* Recent intracranial or intraspinal surgery or trauma (within two months)
* Recent within (2 months) major surgery- Known peptic ulcer or upper gastrointestinal bleeding within the previous 6 month
* Known coagulation anomaly
* Oral anti-coagulant or low molecular weight heparin treatment- Ongoing thrombolytic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-08 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
ST segment regression 1 hour after angioplasty | 1 hour after angioplasty

SECONDARY OUTCOMES:
Major cardiac events at 1 and 6 month | 1 and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Patrick OHLMANN, MD, PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Cardiologie - Hôpital de Hautepierre - 1, Avenue Molière, Strasbourg, France

REFERENCES:
- [Derived] Ohlmann P, Reydel P, Jacquemin L, Adnet F, Wolf O, Bartier JC, Weiss A, Lapostolle F, Gaultier C, Salengro E, Benamer H, Guyon P, Chevalier B, Catan S, Ecollan P, Chouihed T, Angioi M, Zupan M, Bronner F, Bareiss P, Steg G, Montalescot G, Monassier JP, Morel O. Prehospital abciximab in ST-segment elevation myocardial infarction: results of the randomized, double-blind MISTRAL study. Circ Cardiovasc Interv. 2012 Feb 1;5(1):69-76, S1. doi: 10.1161/CIRCINTERVENTIONS.111.961425. Epub 2012 Feb 7. PMID 22319064